CLINICAL TRIAL: NCT00661206
Title: Randomized, Double-Blind, Placebo-controlled Trial of 6 vs. 12 Months Clopidogrel Therapy After Implantation of a Drug-Eluting Stent
Brief Title: Safety and Efficacy of Six Months Dual Antiplatelet Therapy After Drug-Eluting Stenting
Acronym: ISAR-SAFE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A01207
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — Patients on clopidogrel therapy at 6 months after implantation of a drug-eluting stent will be randomized to an additional 6 month period of clopidogrel 75mg per day
  Other Names: Plavix; ACT-Code: B01AC/04
  Arms: Clopidogrel
Drug: Placebo — Patients randomized in this group will receive placebo for 6 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a 6 month duration of clopidogrel therapy after DES implantation is not inferior to that of a 12 month therapy.

DETAILED DESCRIPTION:
Drug elution from stent struts is associated with less smooth muscle cell proliferation and delayed stent strut re-endothelialization. Thus it seems conceivable that a longer duration of dual antiplatelet therapy (aspirin and clopidogrel) after DES implantation is needed. However, no studies have been done to investigate which is the optimal antiplatelet therapy duration after DES implantation. Therefore, the objective of the randomized, double-blind, placebo-controlled ISAR-SAFE study is to evaluate the safety and efficacy of a 6 month versus a 12 month duration of clopidogrel therapy after DES implantation.

Patients on clopidogrel therapy at least 6 months after DES implantation, who do not require a reintervention will be randomized to an additional 6 month period of clopidogrel or placebo. The patients will be followed-up for 9 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients on clopidogrel therapy at 6 months (-1/+2 months) after DES implantation
* Informed, written consent by the patient

Exclusion Criteria:

* Age ≤18 years
* Clinically symptoms, proof of ischemia and/or presence of angiographic lesions requiring revascularization
* Previous stent thrombosis
* DES in left main coronary artery
* ST-elevation and non-ST-elevation myocardial infarction during the last 6 months
* Malignancies or other comorbid conditions with a life expectancy of less than one year or that may result in protocol noncompliance
* Planned major surgery within the next 6 months with the need to discontinue antiplatelet therapy
* Active bleeding; bleeding diathesis; history intracranial bleeding
* Oral anticoagulation therapy with coumadin derivatives
* Known allergy or intolerance to the study medications: aspirin and clopidogrel
* Pregnancy (present, suspected or planned) or positive pregnancy test (In women with childbearing potential a negative pregnancy test is mandatory)
* Patient's inability to fully comply with the study protocol
* Prior enrollment in the same clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4005 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction, stent thrombosis, stroke or TIMI major bleeding. | 9 months after randomization

SECONDARY OUTCOMES:
The individual components of the primary endpoint | 9 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Jurriёn M ten Berg, MD, Principal Investigator — St. Antonius Hospital Nieuwegein, Department of Cardiology
Locations (40):
- University of Florida, Health Science Center - Jacksonville, Jacksonville, Florida, United States
- Spitali Gjerman, Tirana, Albania
- Austria (2):
  - Krankenanstalt Rudolfstiftung, Vienna
  - Wilhelminenspital Wien, Vienna
- University Hospitals Leuven, Leuven, Belgium
- Shenyang Northern Hospital, Shenyang, China
- Aarhus University Hospital, Aarhus, Denmark
- Germany (23):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Charité Berlin, Campus Benjamin Franklin, Berlin
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Universitätsmedizin Göttingen, Göttingen
  - Klinikum Ingolstadt, Ingolstadt
  - MediClin Herzzentrum Lahr/Baden, Lahr
  - Krankenhaus Landshut-Achdorf, Landshut
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Deutsches Herzzentrum München, Munich
  - 1st Medizinische Klinik, Klinikum rechts der Isar, Munich
  - Klinikum Bogenhausen, Munich
  - Klinikum München-Großhadern, München
  - Städtisches Klinikum München-Neuperlach, München
  - Lukaskrankenhaus GmbH, Städtische Kliniken Neuss, Neuss
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinik Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
  - HELIOS Klinikum Wuppertal-Herzzentrum, Wuppertal
- University College Hospital Galway, Galway, Ireland
- Campus Biomedico University of Rome, Rome, Italy
- Japan (2):
  - Tokai University School of Medicine, Isehara
  - Kyoto University Hospital, Kyoto
- Netherlands (4):
  - Catharina Hospital Eindhoven, Eindhoven
  - St. Antonius Hospital Department of Cardiology, Nieuwegein
  - Maasstad Ziekenhuis, Rotterdam
  - Isala klinieken, locatie Weezenlanden, Zwolle
- Auckland City Hospital, Auckland, New Zealand
- Inselspital, Universitätsspital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Schulz-Schupke S, Byrne RA, Ten Berg JM, Neumann FJ, Han Y, Adriaenssens T, Tolg R, Seyfarth M, Maeng M, Zrenner B, Jacobshagen C, Mudra H, von Hodenberg E, Wohrle J, Angiolillo DJ, von Merzljak B, Rifatov N, Kufner S, Morath T, Feuchtenberger A, Ibrahim T, Janssen PW, Valina C, Li Y, Desmet W, Abdel-Wahab M, Tiroch K, Hengstenberg C, Bernlochner I, Fischer M, Schunkert H, Laugwitz KL, Schomig A, Mehilli J, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen: Safety And EFficacy of 6 Months Dual Antiplatelet Therapy After Drug-Eluting Stenting (ISAR-SAFE) Trial Investigators. ISAR-SAFE: a randomized, double-blind, placebo-controlled trial of 6 vs. 12 months of clopidogrel therapy after drug-eluting stenting. Eur Heart J. 2015 May 21;36(20):1252-63. doi: 10.1093/eurheartj/ehu523. Epub 2015 Jan 23. PMID 25616646